CLINICAL TRIAL: NCT06600477
Title: Comparative Randomized, Single Dose, Three-Arm, Parallel Open-Label Study to Characterize the Pharmacokinetics of 7.5 Mg Olanzapine Intranasal Spray and 7.5 Mg Olanzapine Intramuscular Injection After Administration to Healthy Male Adults Under Fasting Conditions
Brief Title: A Study of Olanzapine After Intranasal and Intramuscular Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurelis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OLA-1122-126
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 7.5 mg olanzapine per 100 µL with 0.25% Intravail A3 (Active Comparator): 7.5 mg olanzapine per 100 µL with 0.25% Intravail A3
  Interventions: Drug: olanzapine
- 7.5 mg olanzapine per 100 µL with 0.50% Intravail A3 (Active Comparator): 7.5 mg olanzapine per 100 µL with 0.50% Intravail A3
  Interventions: Drug: olanzapine
- olanzapine intramuscular injection (Active Comparator): 7.5 mg olanzapine per 1.5 ml of reconstituted 5.0 mg/ml solution intramuscular injection
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: olanzapine — 7.5 mg

SUMMARY:
NRL-4, a nasal spray formulation of the atypical antipsychotic olanzapine is being developed by Neurelis Inc. for use as a rescue medication for acute episodes of agitation in schizophrenia, schizoaffective and bipolar I disorder. Also being tested are different concentrations of Intravail A3. Intravail A3 belongs to a class of nonionic surfactants known as alkylglycosides. Alkylglycosides have been extensively studied for their ability to promote increased bioavailability of drugs via the nasal, oral, and ocular routes.

In this study it will be tested if the olanzapine in the two Test products will show comparable pharmacokinetics, safety and tolerability in comparison to the Reference product through the primary pharmacokinetic parameters Cmax, AUC from time 0 to time t and AUC from time 0 to infinity, and safety assessments, including nasal irritation, sedation and pain scales.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18 to 55 years, inclusive.
* Body weight ≥51 kg and ≤111 kg, and body mass index (BMI) range within 18 - 35 kg/m2.
* No clinically significant abnormal findings in the medical and surgical history, on the physical examination, vital sign measurements, electrocardiogram (ECG), or clinical laboratory results during Screening or Admission.
* Written informed consent to participate in the study.
* Capable of returning to study site for all study visits, including the initial confinement period, and willing to comply with all required study procedures.
* Non- or ex-smoker, with ex-smoker defined as someone who completely stopped smoking for at least 6 months before day 1 of the study.
* Sexually active males whose partners are females of childbearing potential must have agreed to use condoms from screening through at least 90 days after administration of study drug and ensured that female partner was using an acceptable form of contraception.

Exclusion Criteria:

* A history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, severe seasonal or non seasonal allergies, nasal polyps or any nasal passage abnormality that could interfere with nasal spray administration, or any other condition which, in the opinion of the Principal Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Treatment with any known enzyme altering drugs such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study drug or during the entire study duration.
* Subjects who have been on an abnormal diet (such as one that severely restricts specific basic food groups [e.g., ketogenic diet], limits calories [e.g., fast], and/or requires the use of daily supplements as a substitute for the foods typically eaten at mealtimes), during the four (4) weeks preceding the study.
* Subjects who donated blood or plasma within 3 months of the first dose of study drug.
* Participation in a bioequivalence study or in a clinical trial with IP administration within 80 days prior to the first dose of study drug.
* Inadequate or difficult venous access that may jeopardize the quality or timing of the PK samples.
* Use of any prescription or over the counter (OTC) medication within 30 days prior to the first dose of study drug or during the study.
* Positive blood screen for HIV, Hepatitis B surface antigen (HbSAg), or Hepatitis C, or a positive screen for alcohol or drugs of abuse.
* History of major depression or suicide attempt, or judged by the investigator as being at significant risk for suicide, violence, or homicide.
* History of postural orthostatic tachycardia syndrome or orthostatic hypotension.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
(1) Bioavailability of test products compared to reference product based on pharmacokinetic parameter of AUC from time 0 to time t | 240 hours
  Characterize the pharmacokinetics of two Test Products (one product, A, is 7.5 mg olanzapine per 100 µL with 0.25% Intravail A3 as absorption enhancer and another product is, B, 7.5 mg olanzapine per 100 µL with 0.50% Intravail A3 as absorption enhancer via nasal spray) relative to Reference Product (C, intramuscular injection) after a single dose of 7.5 mg olanzapine to healthy male adults under fasting conditions.

SECONDARY OUTCOMES:
(2) Bioavailability of test products compared to reference product based on pharmacokinetic parameter of Cmax | 240 hours
  Characterize the pharmacokinetics of two Test Products (one product, A, is 7.5 mg olanzapine per 100 µL with 0.25% Intravail A3 as absorption enhancer and another product is, B, 7.5 mg olanzapine per 100 µL with 0.50% Intravail A3 as absorption enhancer via nasal spray) relative to Reference Product (C, intramuscular injection) after a single dose of 7.5 mg olanzapine to healthy male adults under fasting conditions.
(3) Bioavailability of test products compared to reference product based on pharmacokinetic parameter of AUC from time 0 to infinity | 240 hours
  Characterize the pharmacokinetics of two Test Products (one product, A, is 7.5 mg olanzapine per 100 µL with 0.25% Intravail A3 as absorption enhancer and another product is, B, 7.5 mg olanzapine per 100 µL with 0.50% Intravail A3 as absorption enhancer via nasal spray) relative to Reference Product (C, intramuscular injection) after a single dose of 7.5 mg olanzapine to healthy male adults under fasting conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- International Pharmaceutical Research Center (IPRC) Clinical Site, Amman, Jordan, Jordan

REFERENCES:
- [Derived] Madden S, Citrome L, Correll CU, Shih EK, Lopez-Toledano M, Rabinowicz AL, Carrazana E. A Single-Dose, Randomized, Open-Label, Parallel Design Study to Characterize the Pharmacokinetics of an Investigational Olanzapine Intranasal Spray Compared to a Reference Dose of Olanzapine Intramuscular Injection in Healthy Adult Males. J Clin Psychiatry. 2025 Mar 19;86(2):24m15665. doi: 10.4088/JCP.24m15665. PMID 40117564